CLINICAL TRIAL: NCT05684445
Title: The Effect of Distant Reiki on Pain and Holistic Well-being of Individuals With Phantom Pain After Amputation
Brief Title: The Effect of Distant Reiki on Pain and Holistic Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cemile KÜTMEÇ YILMAZ, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/14-07
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: This study is an experimental one-group pre-test-post-test design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distant reiki group (Experimental): According to Classical Usui Reiki, Reiki II. Remote Reiki will be practiced every day for 10 days by researchers who have completed the Phase 1 training. The time of remote reiki application will be planned by talking with the patient.
  Interventions: Other: Distant reiki group

INTERVENTIONS:
Other: Distant reiki group — According to Classical Usui Reiki, Reiki II. Remote Reiki will be practiced every day for 10 days by researchers who have completed the Phase 1 training. The time of remote reiki application will be planned by talking with the patient.

SUMMARY:
Phantom limb pain is a condition characterized by painful sensations in the missing part of the amputated limb, which reduces the quality of life of the individual. It has been reported that approximately 85% of patients undergoing amputation experience phantom limb pain, and chronic pain is the most common symptom in individuals who have undergone limb amputation. These problems negatively affect individuals physically, mentally and socially and lead to deterioration of holistic well-being. This study will be examined the effect of distant reiki on pain and holistic well-being of ındividuals with phantom pain after amputation.

DETAILED DESCRIPTION:
Phantom limb pain is a condition characterized by painful sensations in the missing part of the amputated limb, which reduces the quality of life of the individual. It has been reported that approximately 85% of patients undergoing amputation experience phantom limb pain, and chronic pain is the most common symptom in individuals who have undergone limb amputation. These problems negatively affect individuals physically, mentally and socially and lead to deterioration of holistic well-being.

Reiki is one of the holistic health practices that is effective in maintaining the balance between body, mind and spirit, which forms the basis of holistic well-being. Reiki, known as an energy-based therapy, helps to rebalance the natural energy flow circulating in the body and to increase the body's self-healing ability, and it prevents or repairs physical, emotional and mental imbalances by regaining the energy we lost in daily life. The purpose of Reiki practice is to promote health and well-being by helping to relax and reduce stress.There is no study in the literature examining the effect of reiki application on phantom pain and holistic well-being.This study was planned to examine the effect of remote reiki applied to individuals with post-amputation phantom pain on pain and holistic well-being.It is thought that it will contribute to the literature in terms of being the first research to be done on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old,
* İndividuals with limb loss and phantom pain
* No communication problem,
* Have the physical and cognitive ability to answer the data collection forms,
* Individuals who have not received body-mind therapy (yoga, reiki, meditation, etc.)

Exclusion Criteria:

* individuals who have done reiki therapy before

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Visual pain Scale | 10 days
  The pain scores of the individuals will be measured after the pre-test and the 10th days using the visual pain scale. Pain score min 1 - max 10. An increase in the score indicates an increase in pain intensity.
Holistic Well-being Scale | 10 days
  Holistic Well-being Scale scores of the individuals will be measured after the pre-test and the 10th days using the Holistic Well-being Scale. The instrument consists of 26 items rated on a 10-point Likert-type scale (1 = strongly disagree to 10 = strongly agree). The scale has no cut-off point.

CONTACTS AND LOCATIONS:
Overall Officials: CEMİLE KÜTMEÇ YILMAZ, Dr., Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Cemile KÜTMEÇ YILMAZ, Merkez, Aksaray
  - Aksaray University Health Science Faculty, Aksaray

IPD SHARING:
Plan to Share IPD: No